CLINICAL TRIAL: NCT02465593
Title: A Phase Ib/II Study of PEP503 (Radioenhancer) With Radiotherapy, in Combination With Concurrent Chemotherapy for Patients With Locally Advanced or Unresectable Rectal Cancer
Brief Title: A Study of PEP503(Radio-enhancer) With Radiotherapy and Chemotherapy for Patients With Rectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PharmaEngine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP503-RC-1001
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Fluorouracil; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEP503+5-FU/capecitabine+Radiotherapy (Experimental): Patients will receive PEP503 given as intratumor injection on Day 1, followed by preoperative radiation therapy.
  Interventions: Drug: PEP503; Drug: 5-fluorouracil; Drug: capecitabine; Procedure: surgical resection; Radiation: Radiotherapy

INTERVENTIONS:
Drug: PEP503 — The volume of PEP503 to be administered is based on the baseline tumor volume of each patient. There will be 4 dose levels in Phase Ib.
  Other Names: NBTXR3
Drug: 5-fluorouracil — 225 mg/m2 a day, 5 days/week for 5 weeks during radiotherapy period
  Other Names: 5-FU
Drug: capecitabine — 825 mg/m2 BID 5 days/week for 5 weeks during the radiotherapy period
  Other Names: Xeloda
Procedure: surgical resection — Approximately 8 weeks after the completion of chemoradiotherapy, surgical resection of the tumor (total mesorectal excision, TME) will be performed once the tumor become resectable.
Radiation: Radiotherapy — Intensity-modulated radiation therapy (IMRT) or intensity modulated arc therapy (IMAT) of 5,000 cGy in 25 fractions (200 cGy/fraction, 5 times/week) to gross tumor and involved nodes and 4,500 cGy in 25 fractions (180 cGy/fraction, 5 times/week) to pelvis, starting at 24 hours after PEP503 injection.

SUMMARY:
This phase Ib/II study is a prospective, open-label, single arm, nonrandomized study of PEP503(radio-enhancer).

There are 2 portions in this study.

* Escalation phase (Part Ib): A 3 + 3 dose escalation study design will be adopted in this phase to identify the recommended injection volume of PEP503 for intratumor injection.
* Expansion phase (Part II): Following the confirmation of the recommended volume of intratumor injection, 18 additional patients will be enrolled at the recommended volume level to evaluate for efficacy.

DETAILED DESCRIPTION:
The target population is composed by patients who have confirmed adenocarcinoma of the rectum which is T3-4, N any, or locally unresectable, with tumor distal margin within 10 cm of the anal verge, with no evidence of distant metastatic disease, ECOG performance 0-1, and adequate bone marrow, renal and hepatic function.

ELIGIBILITY:
Inclusion Criteria

* Histologically proven adenocarcinoma of the rectum which is T3-4, N any, or locally unresectable disease , without evidence of distant metastases (M0)
* Distant border of the tumor must be located ≤ 10 cm from the anal verge
* Staging with MRI, transrectal ultrasound or CT-scan to confirm stage and resectability
* ECOG performance 0 - 1
* Age: 20 - 80 years old
* Adequate bone marrow, renal, and hepatic function as:

  * absolute neutrophil count (ANC) ≥ 1,500/mm3
  * platelet count ≥ 100,000/mm3
  * total bilirubin ≤ 1.5x the upper limit of normal (ULN)
  * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5x ULN
  * alkaline phosphatase (ALP) ≤ 2.5 x ULN
  * calculated creatinine clearance ≥ 50 mL/min, or creatinine within normal range
* All female patients of childbearing potential must have negative urine pregnancy test within the 7 days prior study treatment with PEP503. Patients must agree to use effective contraception during the study

Exclusion Criteria:

* Prior history of pelvic radiation therapy
* Hypersensitivity to fluoropyrimidine
* Uncontrolled serious medical or psychiatric illness
* Myocardial infarction or uncontrolled angor pectoris (angina) within the prior 6 months
* No more than 4 weeks since prior participation in any investigational drug study
* Major surgery within 28 days
* Other malignancy within the past 3 years except effectively treated squamous cell or basal cell skin cancer, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum
* Cardiovascular disease that would preclude study treatment or follow-up
* Informed consent not duly signed and dated to participate in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-06; Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
safety profile /the Dose Limiting Toxicity (DLT) | up to 36 months
  Safety as assess the safety profile and determine the Dose Limiting Toxicity (DLT) of PEP503 given as intratumor injection and activated by external beam radiation, with concurrent chemotherapy in patients with unresectable rectal cancer
the recommended volume (dose) | up to 36 months
  recommended volume (dose) of PEP503 examined by given as intratumor injection and activated by external beam radiation. with concurrent chemotherapy in patients with unresectable rectal cancer
anti-tumor activity | up to 36 months
  Anti-tumor activity as assessed by response rate (RR, as per RECIST 1.1) of PEP503 at the recommended volume given as intratumor injection and activated by external beam radiation, with concurrent chemotherapy in patients with unresectable rectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jwa-Yuan Wang, phD, Principal Investigator — Kaohsiung Municipal United Hospital
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Heald RJ, Ryall RD. Recurrence and survival after total mesorectal excision for rectal cancer. Lancet. 1986 Jun 28;1(8496):1479-82. doi: 10.1016/s0140-6736(86)91510-2. PMID 2425199
- [Background] Colorectal Cancer Collaborative Group. Adjuvant radiotherapy for rectal cancer: a systematic overview of 8,507 patients from 22 randomised trials. Lancet. 2001 Oct 20;358(9290):1291-304. doi: 10.1016/S0140-6736(01)06409-1. PMID 11684209
- [Background] Lubowski DZ. Rectal cancer: the evolving role of adjuvant radiotherapy. ANZ J Surg. 2015 Mar;85(3):99-100. doi: 10.1111/ans.12916. No abstract available. PMID 25732387
- [Background] Tural D, Selcukbiricik F, Yildiz O, Elcin O, Erdamar S, Guney S, Demireli F, Buyukunal E, Serdengecti S. Preoperative versus postoperative chemoradiotherapy in stage T3, N0 rectal cancer. Int J Clin Oncol. 2014 Oct;19(5):889-96. doi: 10.1007/s10147-013-0636-4. Epub 2013 Nov 12. PMID 24218281
- [Result] Nel AE, Madler L, Velegol D, Xia T, Hoek EM, Somasundaran P, Klaessig F, Castranova V, Thompson M. Understanding biophysicochemical interactions at the nano-bio interface. Nat Mater. 2009 Jul;8(7):543-57. doi: 10.1038/nmat2442. Epub 2009 Jun 14. PMID 19525947
- [Derived] Huang CW, Hu HM, Hsu WH, Chen CY, Huang MY, Chen CP, Wei PL, Shen BN, Chang TK, Wang JY. Results of phase Ib/II trial of PEP503 (NBTXR3, radioenhancer) with chemoradiotherapy in patients with rectal cancer. Nanomedicine (Lond). 2025 May;20(9):929-941. doi: 10.1080/17435889.2025.2487411. Epub 2025 Apr 21. PMID 40255171
- [Derived] Huang CW, Hu HM, Hsu WH, Chen CY, Huang MY, Chen CP, Wei PL, Shen BN, Wang JY. A phase Ib/II trial of PEP503 (NBTXR3, radioenhancer) with radiotherapy and chemotherapy in patients with rectal cancer. Nanomedicine (Lond). 2023 Mar;18(6):511-524. doi: 10.2217/nnm-2022-0186. Epub 2023 May 11. PMID 37166053